CLINICAL TRIAL: NCT01050686
Title: Need for Subcutaneous Wound Drains in Ileostomy Reversal
Acronym: DRASTAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Johannes Lauscher, PD Dr. Johannes Lauscher, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA4/120/09
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Presence of Ileostomy
Keywords: ileostomy reversal; subcutaneous drain; hospital stay; postoperative wound infection; patients with elective ileostomy reversal
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- subcutaneous wound drain (Active Comparator): subcutaneous wound drain inserted
  Interventions: Procedure: insertion of subcutaneous wound drain
- no subcutaneous wound drain (Experimental): no subcutaneous wound drain inserted
  Interventions: Procedure: no insertion of subcutaneous wound drain

INTERVENTIONS:
Procedure: insertion of subcutaneous wound drain — after the abdominal fascia is closed and before skin closure, a subcutaneous wound drain is inserted
  Arms: subcutaneous wound drain
Procedure: no insertion of subcutaneous wound drain — closure of abdominal wall and skin without insertion of subcutaneous wound drain
  Arms: no subcutaneous wound drain

SUMMARY:
The purpose of this study is to find out whether the insertion of subcutaneous wound drains has an influence on postoperative hospital stay in ileostomy reversal.

ELIGIBILITY:
Inclusion Criteria:

* elective open reversal of an protective ileostomy

Exclusion Criteria:

* age < 18 years
* missing suitability to comprehend patient information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2010-03; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
length of hospital stay (days) | 3 months postoperatively

SECONDARY OUTCOMES:
surgical site infections | 3 months postoperatively
colonization of abdominal wall with bacteria | 3 months postoperativly
hematomas/ seromas | 3 months postoperatively
postoperative complications | 3 months postoperatively
postoperative pain/ dysaesthesia | 3 months postoperatively
cosmetic result | 3 months postoperatively
postoperative costs | 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Johannes C Lauscher, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Campus Benjamin Franklin; Hindenburgdamm 30, Berlin, State of Berlin, Germany